CLINICAL TRIAL: NCT00659958
Title: Post-authorization, Observational and Prospective Follow up Study to Evaluate Effectiveness and Tolerability of Zonisamide as Adjunctive Therapy in Patients With Partial Onset Seizures Treated With Two Antiepileptic Drugs
Brief Title: ZAGAL Study: Evaluating Effectiveness and Tolerability of Zonisamide as Adjunctive Therapy in Patients With Partial Onset Seizures Treated With Two Antiepileptic Drugs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Eisai Farmacêutica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2090-E044-407
Record Dates: First submitted 2008-04-16; First posted 2008-04-17 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2010-03

CONDITIONS: Epilepsy
Keywords: zonisamide; partial onset seizures; effectiveness; tolerability
MeSH Terms: conditions — Epilepsy | interventions — Zonisamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Zonisamide

INTERVENTIONS:
Drug: Zonisamide — 300 mg tablet. Maintenance dosing period of 12 weeks, at the beginning of which, physicians will decide to keep the 300 mg dose from the titration period, lower it to 200 mg, or take it up to 400 mg.
  Other Names: Zonegran

SUMMARY:
The purpose of this study is to acquire additional information about the appropriate level of dosing of Zonisamide when it is prescribed for patients with partial onset epileptic crisis who are already being treated with two other antiepileptic drugs.

DETAILED DESCRIPTION:
Patients from both sexes, 18 to 65 years of age, diagnosed with simple or complex partial onset epileptic crisis defined according to the International League Against Epilepsy (ILAE) criteria, with a minimum of two seizures within the 4 previous weeks, a stable treatment with two antiepileptic drugs for at least 12 weeks, and capable and willing to give their informed consent, will be included in the study.

To these patients, physicians will prescribe zonisamide in the following manner: Titration period of 12 weeks, at the end of which all patients must be taking 300 mg. Maintenance doses period of 12 weeks, at the beginning of which, physicians will decide to keep the 300 mg dose from the titration period, lower it to 200 mg, or take it up to 400 mg. Six weeks later within this period, a decision will be made to raise the 400 mg doses up to 500 mg if considered necessary and tolerable.

Drugs will be prescribed by the physician and purchased by the patient.

ELIGIBILITY:
Inclusion Criteria:

Patients from both sexes, 18 to 65 years of age, diagnosed with simple or complex partial onset epileptic seizures defined according to the International League Against Epilepsy (ILAE) criteria, with a minimum of two crises within the 4 previous weeks, a stable treatment with two antiepileptic drugs for at least 12 weeks and capable and willing to give their informed consent, will be included.

Exclusion Criteria:

Those who do not fulfill the Inclusion requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Frequency of seizures. | Evaluations will be done at the beginning of the study (enrollment visit) and then one more time when 24 weeks had passed.

SECONDARY OUTCOMES:
Quality of life, tolerability. | Quality of Life evaluations will be done at the beginning of the study (enrollment visit) and then one more time when 24 weeks have passed. Tolerability will be assessed at the beginning of the study (enrollment visit) and at 12, 18, and 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus De Rosendo, Study Chair — EISAI Farmaceutica S.A. Head of Medical Department
Locations (11):
- Spain (11):
  - Complejo Hospitalario Universitario 'Juan Canalejo', A Coruña, Galicia
  - C.H. A. Marcide Profesor Novoa Santos, Ferrol, Galicia
  - Centro Sanitario Complexo Hospitalario "XERAL-CALDE", Lugo, Galicia
  - Hospital Comarcal de Monforte, Lugo, Galicia
  - Centro Sanitario Hospital Da Costa de Burela, Lugo, Galicia
  - Complejo Hospitalario de Ourense, Ourense, Galicia
  - Complejo Hospitalario de Pontevedra, Pontevedra, Galicia
  - Complejo Hospitalario Universitario Santiago de Compostela, Santiago de Compostela, Galicia
  - Complejo Hospitalario Universitario de Vigo (CHUVI), Hospital Meixoeiro, Vigo, Galicia
  - Hospital Povisa, Vigo, Galicia
  - Complejo Hospitalario Universitario de Vigo (CHUVI), Hospital Xeral-Cies, Vigo, Galicia